CLINICAL TRIAL: NCT02841735
Title: Young Adult Naturalistic Alcohol Study (YANAS) Using Smartphone Technology in a Simulated Laboratory Environment
Status: Terminated | Type: Observational
Why Stopped: Protocol expired with IRB.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201500990; ID00004419 (Other Grant/Funding Number: Health & Human Performance)
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Alcohol Use; Alcohol Drinking; Drinking Behavior
Keywords: brief intervention; web-based interventions; harm reduction; young adult; college student
MeSH Terms: conditions — Alcohol Drinking; Drinking Behavior; Harm Reduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Smartphone breathalyzer device & app: This is a small device that attaches to a smartphone with an accompanying app that produces accurate breath alcohol readings when a user blows into a small tube attached to the device. Participants randomized to this study condition will have the opportunity to use this device and app during an alcohol drinking session in a simulated laboratory.
  Interventions: Device: Smartphone breathalyzer device/app use
- BAC estimator app: This is an app that produces estimated blood alcohol content (eBAC) readings based on sex, weight, number of drinks and time taken to consume drinks. Participants randomized to this study condition will have the opportunity to use this app during an alcohol drinking session in a simulated laboratory.
  Interventions: Device: BAC estimator app use
- Text Messaging: A procedure whereby one sends a text message to the phone one is using after each alcoholic drink. Participants randomized to this study condition will have the opportunity to the text messaging procedure during an alcohol drinking session in a simulated laboratory.
  Interventions: Device: Text messaging procedure

INTERVENTIONS:
Device: Smartphone breathalyzer device/app use — Participants randomized to this condition will be able to blow into the smartphone breathalyzer after consuming each alcoholic drink, which produces an accurate breath alcohol reading on the app. These breath alcohol readings may inform participants' subsequent decisions regarding drinking.
  Groups: Smartphone breathalyzer device & app
Device: BAC estimator app use — Participants randomized to this condition will be able to make an entry into the BAC estimator app after consuming each alcoholic drink, which produces an estimated blood alcohol concentration based on the individual's sex, weight, number of alcoholic drinks and time spent drinking alcohol. These estimated blood alcohol concentrations may inform participants' subsequent decisions regarding drinking.
  Groups: BAC estimator app
Device: Text messaging procedure — Participants randomized to this condition will be instructed to send a text to a smartphone they will use for the study after each alcoholic drink. A consideration of the number of texts sent may inform participants' subsequent decisions regarding drinking.
  Groups: Text Messaging

SUMMARY:
It is important to explore use of technology to reduce drinking. The purpose of this research study is to compare different types of mobile technology for their effects on alcohol drinking and ratings of usability among young adults.This study will be conducted in four phases: a web-based screening assessment; brief appointment on the day of the alcohol drinking session; alcohol drinking session; and a follow-up appointment. Participation in this study will last approximately two months.

ELIGIBILITY:
Inclusion Criteria:

* Be able to read English and complete assessments
* Drink alcohol regularly

Exclusion Criteria:

* Test positive on a urine test for use of certain illegal drugs
* Undergraduate student enrolled in the University of Florida
* Graduate students from the College of Health and Human Performance at the University of Florida
* Pregnant, or breast feeding

Ages: 21 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Interested individuals will contact the study by telephone or by email or will go directly to the study's information page located at www.yanasinfo.org.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2016-07; Primary Completion 2018-02-03 (Actual); Study Completion 2018-02-03 (Actual)

PRIMARY OUTCOMES:
Quantity of alcohol consumption | During an alcohol drinking session
  Compare forms of mobile technology for their effects on alcohol consumption

CONTACTS AND LOCATIONS:
Overall Officials: Robert F. Leeman, Ph.D., Principal Investigator — University of Florida
Locations (1):
- Department of Health Education and Behavior, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No